CLINICAL TRIAL: NCT07160530
Title: Cluster Randomized Controlled Trial of a Multilevel Rural Community Engagement Model for Improving Children's Dietary Intake in Family Child Care Homes
Brief Title: Healthy Children, Healthy Communities: Effectiveness of a Multilevel Rural Community Engagement Model for Improving Children's Dietary Intake in Family Child Care Homes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska Lincoln (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: UNL-00024617
Record Dates: First submitted 2025-07-10; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Childhood Obesity Pevention; Diet Quality; Feeding Behaviors; Health Behavior Change; Rural Health
Keywords: Rural population; Feeding Behavior; Child Care; Child Feeding; Carotenoids; Body Mass Index
MeSH Terms: conditions — Feeding Behavior | interventions — Eating

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 2. Better Kid Care (Active Comparator): Arm 2: Rural family childcare home providers receive 10 online modules about general childcare topics unrelated to nutrition, including child development, block play, oral health, supervising children, and managing a family childcare home through the Better Kid Care platform.
  Interventions: Behavioral: Better Kid Care
- Arm 1: EAT Family Style (Experimental): Arm 1: Rural family childcare home providers receive 7 online modules on responsive feeding practices over 16 weeks, plus 7 individual coaching sessions via Zoom with Extension agents. Providers record mealtime videos for personalized feedback, engage in goal-setting and action planning, and receive printed materials and conversation cards.
  Interventions: Behavioral: EAT Family Style

INTERVENTIONS:
Behavioral: EAT Family Style — Rural family childcare home providers receive 7 online modules on responsive feeding practices over 16 weeks, plus 7 individual coaching sessions via Zoom with Extension agents. Providers record mealtime videos for personalized feedback, engage in goal-setting and action planning, and receive printed materials and conversation cards.
  Other Names: EAT for Prevention
  Arms: Arm 1: EAT Family Style
Behavioral: Better Kid Care — Rural family childcare home providers receive 10 online modules about general childcare topics unrelated to nutrition, including child development, block play, oral health, supervising children, and managing a family childcare home through the Better Kid Care platform.
  Arms: Arm 2. Better Kid Care

SUMMARY:
The purpose of this study is to find out whether a program called "Healthy Children, Healthy Communities" can help young children in rural areas eat healthier and improve their health. The study focuses on children ages 3 to 5 who attend family childcare homes in rural communities.

The main goal is to see if the program can:

Help children eat healthier foods, like more fruits and vegetables.

Support childcare providers in using positive mealtime practices that encourage healthy eating.

The study will involve about 120 licensed family childcare providers in rural areas who participate in the Child and Adult Care Food Program (CACFP), along with about 240 children they care for.

Childcare providers will be randomly placed into one of two groups:

EAT Family Style Group (Intervention Group):

Complete 7 online training modules over 16 weeks about healthy mealtime practices.

Join 7 individual coaching sessions on Zoom.

Record short videos of their mealtimes to get personalized feedback from a coach.

Work with a coach to set goals and make plans to improve mealtimes.

Receive printed materials and conversation cards to use during meals.

Some providers may join Zoom interviews to share their experiences.

Better Kid Care Group (Comparison Group):

Complete 10 online modules about general childcare topics like child development, oral health, play, and managing a childcare home.

For both groups, the research team will:

Ask providers to fill out online surveys about how mealtimes work in their childcare homes.

Visit the childcare homes to observe and record children's mealtimes on two days at each data collection point.

Measure the height and weight of participating children.

Use a painless skin scanner (Veggie Meter) to check how many fruits and vegetables children have been eating.

Ask providers to complete surveys about the children's eating habits.

The study focuses on rural, low-income communities, where children are at higher risk of having poor diets and obesity compared to children in urban areas. Information will be collected at the start of the study, after 16 weeks, and again after 24 weeks to see if there are lasting changes.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the effectiveness of a multilevel rural community engagement model in:

1. improving children's dietary intake, and
2. enhancing providers' feeding practices, within rural family childcare homes, using a cluster randomized controlled trial design.

Secondary objectives are to assess within these family childcare homes:

1. child BMI z-scores and skin carotenoid levels (as a biomarker of fruit and vegetable intake), and
2. the mealtime emotional climate.

This cluster randomized controlled trial uses the family childcare home as the unit of randomization (i.e., clusters), with both children and providers nested within each family childcare home.

ELIGIBILITY:
Inclusion Criteria:

FCCH Settings:

* Licensed family child care home-based early child care and education settings
* Located in Nebraska (with potential expansion to Iowa, Kansas, South Dakota, Oklahoma, Illinois, and/or Northwest Missouri if needed)
* Participate in the Child and Adult Care Food Program (CACFP)
* Care for at least 2 preschool-aged non-sibling children (3-5 years old) without feeding disorders or developmental delays
* Provide meals and snacks to attending children
* Located in a county designated as nonmetropolitan based on the 2023 Rural-Urban Continuum Codes (RUCC)

FCCH Providers:

* Currently caring for at least two 3-5 year old non-sibling children who do not have dietary restrictions or feeding disorders that impact how they eat
* Present with children during meals and snacks
* Over the age of 19 years
* Have not participated in this study before

Children:

* Between 3 to 5 years old
* No dietary restrictions or feeding disorder that impact how they eat (lactose intolerance, egg/nut allergies, or vegetarian diet are acceptable)
* Typically developing children (no diagnosis of developmental delays as identified by childcare providers)
* Have a parent or guardian 19 years of age or older to consent for them

Exclusion Criteria:

FCCH Providers:

* FCCH provider closes the business
* FCCH provider stops serving meals to children
* FCCH provider discontinues participation in CACFP and no longer adheres to CACFP meal pattern requirements
* FCCH provider loses all eligible study children due to children leaving care, developing developmental delays or feeding disorders, or other reasons making them ineligible

Children:

* Diagnosis of dietary restrictions or feeding disorder that impact how they eat (soft diet requirements or difficulty swallowing that impacts how they eat)
* Diagnosis of developmental delays
* A sibling of a participating child (only one 3-5 year old child per family eligible)

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2025-10-07 (Estimated); Primary Completion 2028-12-20 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in children's observed combined fruit and vegetable consumption [16 weeks] | From baseline to 16 weeks post-intervention
  Children's fruit and vegetable consumption (servings/day) will be assessed by trained research staff observing two consecutive days of meals and snacks in family child care homes (FCCHs), following the Dietary Observation in Child Care (DOCC) protocol, which allows one observer to record intake for up to three children with minimal disruption.
  Data will be entered into the Nutrition Data System for Research (NDSR) to convert observed foods into nutrient and food group values.
  Fruit and vegetable intake will be quantified using MyPlate categories and compared to Dietary Guidelines for Americans to determine each child's two-day average intake.
Change in children's observed combined fruit and vegetable consumption [24 weeks] | From baseline to 24 weeks post-intervention
  Children's fruit and vegetable consumption (servings/day) will be assessed by trained research staff observing two consecutive days of meals and snacks in family child care homes (FCCHs), following the Dietary Observation in Child Care (DOCC) protocol, which allows one observer to record intake for up to three children with minimal disruption.
  Data will be entered into the Nutrition Data System for Research (NDSR) to convert observed foods into nutrient and food group values.
  Fruit and vegetable intake will be quantified using MyPlate categories and compared to Dietary Guidelines for Americans to determine each child's two-day average intake.

SECONDARY OUTCOMES:
Change in children's observed diet quality, measured by the Healthy Eating Index-2020 (HEI-2020) (16 weeks) | From baseline to 16 weeks post-intervention
  Children's dietary intake will be assessed by trained research staff observing two days of meals and snacks in family child care homes (FCCHs), following the Dietary Observation in Child Care (DOCC) protocol, which allows one observer to record intake for up to three children with minimal disruption. Data will be entered into the Nutrition Data System for Research (NDSR) to convert observed foods into nutrient and food group values. Diet quality will be measured with the Healthy Eating Index-2020 (HEI-2020), ranging from 0-100, where higher scores reflect better diet quality. Average HEI-2020 scores will be calculated per child, standardized per 1,000 kcal, and aggregated at the FCCH level.
Change in children's observed diet quality, measured by the Healthy Eating Index-2020 (HEI-2020) (24 weeks) | From baseline to 24 weeks follow-up
  Children's dietary intake will be assessed by trained research staff observing two days of meals and snacks in family child care homes (FCCHs), following the Dietary Observation in Child Care (DOCC) protocol, which allows one observer to record intake for up to three children with minimal disruption. Data will be entered into the Nutrition Data System for Research (NDSR) to convert observed foods into nutrient and food group values. Diet quality will be measured with the Healthy Eating Index-2020 (HEI-2020), ranging from 0-100, where higher scores reflect better diet quality. Average HEI-2020 scores will be calculated per child, standardized per 1,000 kcal, and aggregated at the FCCH level.
Change in the observed mealtime emotional climate | From baseline to 16 weeks post-intervention and 24-week follow-up
  Mealtime emotional climate refers to the quality of interpersonal interactions between the provider and children during mealtime. We will record lunchtime videos during baseline, post and follow-up to assess MEC coded by the Mealtime Emotional Climate in Child Care Observational Scales , which includes two higher-level constructs: positive and negative MEC.
Change in family childcare home providers observed responsive feeding practices (16 weeks) | From baseline to 16 weeks post-intervention
  Providers' observed responsive feeding practices. The research team will record lunchtime videos before and after the intervention and follow-up; these videos will be coded using the Mealtime Observation in Child Care Checklist. These responsive feeding practices are focused on improving mealtime structure and providing developmentally appropriate support for children's autonomy.
Change in family childcare home providers observed responsive feeding practices (24 weeks) | From baseline to 24 weeks follow-up
  Providers' observed feeding practices. The research team will record lunchtime videos before and after the intervention and follow-up; these videos will be coded using the Mealtime Observation in Child Care Checklist. These responsive feeding practices are focused on improving mealtime structure and providing developmentally appropriate support for children's autonomy.
Change in family childcare home providers' self-reported responsive feeding practices (16 weeks) | From baseline to 16 weeks post-intervention
  Providers' self-reported feeding practices. All FCCH providers will complete a 30- 45-minute online survey on Qualtrics before, after, and during follow-up data collection to to measure providers' responsive feeding practices. These practices are focused on improving mealtime structure and providing developmentally appropriate support for children's autonomy during mealtimes.
Change in family childcare home providers' self-reported responsive feeding practices (24 weeks) | From baseline to 24-week follow-up
  Providers' self-reported responsive feeding practices. All FCCH providers will complete a 30- 45-minute online survey on Qualtrics before, after, and during follow-up data collection to to measure providers' responsive feeding practices. These practices are focused on improving mealtime structure and providing developmentally appropriate support for children's autonomy during mealtimes.
Change in family childcare home providers observed controlling feeding practices (16 weeks) | From baseline to 16 weeks post-intervention
  Providers' observed controlling feeding practices (e.g. pressure to eat, offering food as reward). The research team will record lunchtime videos before and after the intervention and follow-up; these videos will be coded using the Mealtime Observation in Child Care Checklist.
Change in family childcare home providers observed controlling feeding practices (24 weeks) | From baseline to 24 weeks follow-up
  Providers' observed controlling feeding practices (e.g. pressure to eat, offering food as reward). The research team will record lunchtime videos before and after the intervention and follow-up; these videos will be coded using the Mealtime Observation in Child Care Checklist.
Change in family childcare home providers' self-reported controlling feeding practices (16 weeks) | From baseline to 16 weeks post-intervention
  Providers' self-reported controlling feeding practices (e.g. pressure to eat, offering food as reward). All FCCH providers will complete a 30- 45-minute online survey on Qualtrics before, after, and during follow-up data collection to to measure providers' controlling feeding practices.
Change in family childcare home providers' self-reported controlling feeding practices (24 weeks) | From baseline to 24 weeks follow-up
  Providers' self-reported controlling feeding practices (e.g. pressure to eat, offering food as reward). All FCCH providers will complete a 30- 45-minute online survey on Qualtrics before, after, and during follow-up data collection to to measure providers' controlling feeding practices.

OTHER OUTCOMES:
Change in children's skin carotenoids (16 weeks) | From baseline to 16 weeks post-intervention
  The Veggie Meter device (Longevity Link Corp., Utah)will provide an objective, non-invasive, and quick measure reflecting fruit and vegetable intake at all three study timepoints. The device uses reflection spectroscopy to detect carotenoid levels in human skin, has been validated against dietary intake in diverse groups of adults and children and also assess changes over time.
Change in children's skin carotenoids (24 weeks) | From baseline to 24-week follow-up
  The Veggie Meter device (Longevity Link Corp., Utah)will provide an objective, non-invasive, and quick measure reflecting fruit and vegetable intake at all three study timepoints. The device uses reflection spectroscopy to detect carotenoid levels in human skin, has been validated against dietary intake in diverse groups of adults and children and also assess changes over time.
Change in children's measured BMI z-score (16 weeks) | From baseline to 16 weeks post-intervention
  Children's standing height (in meters) will be measured using a portable stadiometer, and weight (in kg) will be measured using a calibrated digital scale in the FCCH setting, following a standard protocol. Height-weight measurements will be aggregated to arrive at BMI z-score (e.g., weight and height will be combined to report BMI in kg/m^2 and then calculate the BMI z-score).
Change in children's measured BMI z-score (24 weeks) | From baseline to 24-week follow-up
  Children's standing height (in meters) will be measured using a portable stadiometer, and weight (in kg) will be measured using a calibrated digital scale in the FCCH setting, following a standard protocol. Height-weight measurements will be aggregated to arrive at BMI z-score (e.g., weight and height will be combined to report BMI in kg/m^2 and then calculate the BMI z-score).

CONTACTS AND LOCATIONS:
Overall Officials: Dipti Dev, PhD, Principal Investigator — University of Nebraska Lincoln
Locations (1):
- University of Nebraska Lincoln, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to make IPD and related data dictionaries available. All collected individual participant data that underlies results in publications will be shared after being fully de-identified. This includes child dietary intake, anthropometric, skin carotenoid data, provider feeding practices surveys, and demographic information. Data will be available through the NICHD DASH controlled-access repository with proper plans and safeguards for privacy protection.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will become available as soon as the dataset is cleaned and prior to the time of publication or the end of the funding period, whichever comes first. Data will be permanently archived and maintained through the NICHD DASH repository for long-term access and preservation, following NIH data sharing policies.
Access Criteria: Access will be provided through NICHD's DASH controlled-access repository to identity-verified researchers for scientifically and ethically appropriate uses. The NICHD DASH Data Access Committee reviews all access requests to ensure proposed use does not conflict with research data use limitations. Requesters must establish a Data Use Agreement outlining expectations for appropriate use of DASH data.
URL: https://dash.nichd.nih.gov/